CLINICAL TRIAL: NCT05077761
Title: High-intensity Laser Therapy on Hamstring Muscle Length Among Young Adults
Brief Title: Laser Therapy on Hamstring Muscle Among Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Asir John Samuel, Associate Professor, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1269-9595
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Muscle Tightness
Keywords: Flexibility; Hamstring; Laser therapy; Young adults

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity laser therapy (Experimental): 77 participants will receive active high-intensity laser therapy interventions on hamstring muscle to improve the flexibility of muscle
  Interventions: Device: Active High-intensity laser therapy
- Sham High-intensity laser therapy (Sham Comparator): 77 participants will receive sham high-intensity laser therapy on hamstring muscle
  Interventions: Device: Sham High-intensity laser therapy

INTERVENTIONS:
Device: Active High-intensity laser therapy — High-intensity laser therapy will be used in the contact method, with the laser beam irradiated over the hamstring muscle. Dosage and parameters for the laser will be calculated.
  Parameters-
  1. Wavelength- 980 nm
  2. Intensity/Power density- 3W/cm2
  3. Emission mode- Continuous Emission
  4. Energy (Joules)- 490 J
  5. Irradiation time- 70 Sec on each point
  6. Peak power- 15 Watt
  7. Irradiation points- 09
  Arms: High-intensity laser therapy
Device: Sham High-intensity laser therapy — Sham High-intensity laser therapy will be used in the contact method, without the laser beam irradiation over the hamstring muscle.
  Arms: Sham High-intensity laser therapy

SUMMARY:
A total of 154 healthy young individuals will be recruited by purposive sampling method to participate in a randomized, single-blinded, sham-controlled study. Recruited participants will be randomly dividing into two groups, the Active high-intensity laser therapy (a-HILT) group, and the Sham high-intensity laser therapy (s-HILT) group. The treatment duration will be 10 minutes per session on both lower limbs for each day for 3 days/week for 2 weeks. Hamstring muscle length will be assessed at baseline, end of the 2-week post-intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic young adults
* Both gender
* Tightness of hamstring muscles

Exclusion Criteria:

* Any other musculoskeletal disorder
* Any disc pathology
* Any nerve root irritation
* Any surgical history or trauma
* Malignancy
* Pregnancy
* Sensory dysfunctions
* Cardiac pacemaker

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-08-19 (Actual); Study Completion 2023-10-09 (Actual)

PRIMARY OUTCOMES:
Active Knee Extension Test | Changes will be measured at baseline, end of two week post intervention
  Active knee extension test (AKET) is most reliable method to assess the hamstring tightness.
Sit and toe touch test | Changes will be measured at baseline, end of two week post intervention
  Sit and toe touch test is used to assess the hamstring flexibility

CONTACTS AND LOCATIONS:
Overall Officials: Adarsh K Srivastav, PhD Scholar, Principal Investigator — MMIPR, MM(DU); Asir J Samuel, PhD, Study Director — MMIPR, MM(DU)
Locations (1):
- Maharishi Markandeshwar (M.M) Hospital, Mullana, Ambala, Haryana, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cejudo A, Centenera-Centenera JM, Santonja-Medina F. The Potential Role of Hamstring Extensibility on Sagittal Pelvic Tilt, Sagittal Spinal Curves and Recurrent Low Back Pain in Team Sports Players: A Gender Perspective Analysis. Int J Environ Res Public Health. 2021 Aug 16;18(16):8654. doi: 10.3390/ijerph18168654. PMID 34444402
- [Background] Jozwiak M, Pietrzak S, Tobjasz F. The epidemiology and clinical manifestations of hamstring muscle and plantar foot flexor shortening. Dev Med Child Neurol. 1997 Jul;39(7):481-3. doi: 10.1111/j.1469-8749.1997.tb07468.x. PMID 9285439
- [Background] Medeiros DM, Aimi M, Vaz MA, Baroni BM. Effects of low-level laser therapy on hamstring strain injury rehabilitation: A randomized controlled trial. Phys Ther Sport. 2020 Mar;42:124-130. doi: 10.1016/j.ptsp.2020.01.006. Epub 2020 Jan 10. PMID 31991284
- [Background] Dornelles MP, Fritsch CG, Sonda FC, Johnson DS, Leal-Junior ECP, Vaz MA, Baroni BM. Photobiomodulation therapy as a tool to prevent hamstring strain injuries by reducing soccer-induced fatigue on hamstring muscles. Lasers Med Sci. 2019 Aug;34(6):1177-1184. doi: 10.1007/s10103-018-02709-w. Epub 2019 Jan 3. PMID 30607719
- [Background] Hughes T, Callaghan M. BET 2: LASER THERAPY IN THE TREATMENT OF ACUTE HAMSTRING MUSCLE INJURIES. Emerg Med J. 2017 Apr;34(4):266. doi: 10.1136/emermed-2017-206665.2. PMID 28341795
- [Background] Ramos GA, Arliani GG, Astur DC, Pochini AC, Ejnisman B, Cohen M. Rehabilitation of hamstring muscle injuries: a literature review. Rev Bras Ortop. 2016 Dec 15;52(1):11-16. doi: 10.1016/j.rboe.2016.12.002. eCollection 2017 Jan-Feb. PMID 28194375